CLINICAL TRIAL: NCT01538784
Title: A Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of YF476, a Novel, Potent and Selective Gastrin/Cholecystokinin-B Antagonist, in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Doses of YF476, a Gastrin Antagonist, in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 96-001
Record Dates: First submitted 2012-02-15; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Reflux Oesophagitis
Keywords: YF476; gastrin receptor antagonist; gastric pH; healthy subjects
MeSH Terms: conditions — Esophagitis, Peptic | interventions — YF 476

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: YF476 — Two groups of six subjects received single rising oral doses of YF476 capsules or matching placebo. Each subject received 2 doses of YF476 and 1 dose of placebo. 4 subjects received active and 2 placebo at each dose level, as follows:
  Group A YF476 0.5, 25 and 100mg by mouth Group B YF476 5.0, 50 and 100mg by mouth
  Groups A & B were dosed alternately, at weekly intervals

SUMMARY:
The objectives of the study were:

* To assess the safety, tolerability and pharmacokinetics of YF476 in healthy volunteers.
* To select a dose or doses of YF476 for detailed pharmacodynamic studies in healthy volunteers.

DETAILED DESCRIPTION:
YF476 is clearly a potent and selective gastrin/CCK-B antagonist and should inhibit basal and meal-stimulated gastric acid secretion and enhance gastric emptying of a liquid meal in man. Therefore YF476 might benefit patients with reflux oesophagitis. The compound has been remarkably well tolerated in animal toxicity studies at doses well in excess of the projected therapeutic dose in patients, and merits first administration to healthy volunteers. That study using the oral route of administration is described here. Extrapolation from data obtained with pentagastrin in animals suggest that single doses of less than 1mg of YF476 should be active in man. However, extrapolation from data obtained in comparative studies with the H2-antagonists and with omeprazole in animals suggest that the therapeutic dose in patients with reflux oesophagitis will be larger, in the region of 10mg. A range of single doses will be used in this study. The maximum dose will be 10 times more than the expected therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and aged 18-45 years.
* No clinically relevant abnormal findings in the clinical history or physical examination at the screening assessment which could interfere with the objectives of the study or make the subject's participation hazardous.
* No clinically relevant abnormal laboratory values at the screening evaluation (Attachment 2).
* A normal ECG at the screening examination.
* A body mass index (Quetelet index) in the range 19-30:
* Body Mass Index = weight [kg]_ height [m]2
* Normal blood pressure and heart rate at the screening examination, i.e. BP 90-150mmHg systolic, 40-95mmHg diastolic; heart rate 40-100 beats/min in seated position.
* Subjects must be of sufficient intelligence to understand the nature of the study and any hazards of their participation in it. They must be able to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study.
* Subjects must give their written consent to participate after reading the Information-for-Volunteers Leaflet and Consent Form, and after having the opportunity to discuss the study with the Investigator or his deputy.

Exclusion Criteria:

* Clinically relevant abnormal history or physical findings at the screening assessment, which could interfere with the objectives of the study or the safety of the subject's participation.
* Clinically relevant abnormalities of laboratory values or ECG at screening evaluation.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate subject's participation in the study or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease or history of any psychotic mental illness.
* Participation in other clinical studies of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or intake of more than 40 units of alcohol weekly.
* Loss of more than 400ml blood during the 3 months before the study, e.g. as a blood donor.
* Use of prescription medication during 30 days before the study.
* Use of an over-the-counter medicine during 7 days before the study
* Blood pressure or heart rate outside those values specified under inclusion criterion (f).
* Possibility that the subject will not cooperate with the requirements of the protocol.
* Evidence of drug abuse on urine testing at study entry.
* Positive test for hepatitis B or C or HIV 1 & 2.
* High risk of hepatitis or HIV infection.
* History of severe allergic disease.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 1996-05; Primary Completion 1996-06 (Actual); Study Completion 1996-06 (Actual)

PRIMARY OUTCOMES:
Clinically relevant changes from baseline in safety assessments | 6 weeks
  Physical examination, ECG and safety tests of blood and urine at screening and at 24 hours and 7 days after dosing. ECG, blood pressure and heart rate during study period.
Numbers of adverse events | 6 weeks
  Adverse events during study period and at follow-up.
Pharmacokinetic parameters: Cmax, Tmax, AUC 0-24 h, T1/2 | 6 weeks
  Blood samples (10 mL) for assay of YF476 at 0, 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hours after dosing.
  Urine collection: 0-6, 6-12 and 12-24 hours after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J Boyce, FRCP FFPM, Study Director — Trio Medicines Limited
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Derived] Boyce M, David O, Darwin K, Mitchell T, Johnston A, Warrington S. Single oral doses of netazepide (YF476), a gastrin receptor antagonist, cause dose-dependent, sustained increases in gastric pH compared with placebo and ranitidine in healthy subjects. Aliment Pharmacol Ther. 2012 Jul;36(2):181-9. doi: 10.1111/j.1365-2036.2012.05143.x. Epub 2012 May 20. PMID 22607579